CLINICAL TRIAL: NCT04564924
Title: To Investigate the Bone and Muscle Abnormalities in Patients With Chronic Kidney Disease Compared to Healthy Volunteers With MRI
Brief Title: To Investigate the Bone and Muscle Abnormalities in Patients With Chronic Kidney Disease With MRI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, yan Xiong, PhD, Tongji Hospital
Other Study IDs: S094
Record Dates: First submitted 2020-09-14; First posted 2020-09-25 (Actual); Last update posted 2020-09-25 (Actual); Status verified 2020-09

CONDITIONS: Chronic Kidney Disease-Mineral and Bone Disorder
MeSH Terms: conditions — Chronic Kidney Disease-Mineral and Bone Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine, serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- MRI & DXA patients: No intervention
  Interventions: Radiation: DXA
- MRI & DXA volunteers: No intervention
  Interventions: Radiation: DXA

INTERVENTIONS:
Radiation: DXA — Bone mineral density was examined in all cases and controls

SUMMARY:
Patients with chronic kidney disease (CKD) have a higher risk of fractures than those without. The purpose of this study is to develop a non-invasive Magnetic resonance imaging (MRI) method that can improve fracture risk prediction and provide early diagnosis for bone abnormalities in patients with CKD.

DETAILED DESCRIPTION:
Chronic Kidney Disease-Mineral and Bone Disorder (MBD） is a common complication of chronic kidney disease (CKD), which may lead to defective mineralization, altered bone morphology, and/or bone turnover. Animal research found that bone changes occur even in the early stage of CKD , and with CKD progression, the patient may show symptoms such as bone pain, joint pain, bone deformation, and even spontaneous fractures.

Despite significant advances in understanding bone disease in CKD, most clinical and biochemical targets used in clinical practice remain controversial, resulting in an undermanagement of bone fragility.Our ability to diagnose CKD-MBD and to initiate strategies that could prevent fractures remains limited by the lack of accurate and noninvasive diagnostic tools.

The purpose of this study is to develop a non-invasive method that can improve fracture risk prediction and provide early diagnosis for bone abnormalities in patients with CKD.

ELIGIBILITY:
Inclusion Criteria:

CKD patients aged 18-70 years with free movement

-

Exclusion Criteria:

1. The following diseases: rickets, osteomalacia, Paget's disease, acromegaly, scurvy (vitamin C deficiency), hyperthyroidism, history of malignant tumors, received radiotherapy and chemotherapy, fractures within 6 months, lumbar and calf trauma surgery, scoliosis, rheumatic immunity disease, anorexia nervosa, motor neuron disease
2. Treated with the following drugs within two years:

   A) Bisphosphonates: Alendronate , etidronate , Ibandronate, rithiadronate, and zoledronate B) Steroid hormones: estrogen replacement agents , isoflavone derivatives , estrogen, progesterone C) Oral glucocorticoids: prednisone , Prednisone D) Salmon calcitonin
3. MRI contraindications: Intra Uterine Device(iUD), pacemaker, cochlear implant, claustrophobia, etc -

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subject group:Hospitalized patients in department of Nephrology, Tongji Hospital, Qiaokou District, Wuhan, Hubei, China control group:social recruitment
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-09-02 (Actual); Primary Completion 2021-09-30 (Estimated); Study Completion 2022-01-30 (Estimated)

PRIMARY OUTCOMES:
Magnetic resonance examination for general diagnosis：routine imaging sequences | 12 months
  All MRI imaging was performed on a clinical 3.0 T General Electric(GE) MR scanner on the lumbar spine and lower legs of both experimental group and control group.
Magnetic resonance examination to measure tissue diffusion and perfusion：DWI-related sequence | 12 months
  All MRI imaging was performed on a clinical 3.0 T General Electric(GE) MR scanner on the lumbar spine and lower legs of both experimental group and control group.And the full abbreviation of the above sequence:Diffusion Weighted Imaging(DWI)-related sequence
Magnetic resonance examination to measure material changes in tissue：CEST | 12 months
  All MRI imaging was performed on a clinical 3.0 T General Electric(GE) MR scanner on the lumbar spine and lower legs of both experimental group and control group.And the full abbreviation of the above sequence: chemical exchange saturation transfer(CEST)
Magnetic resonance examination to measure the fat content of tissues：IDEAL- IQ | 12 months
  All MRI imaging was performed on a clinical 3.0 T General Electric(GE) MR scanner on the lumbar spine and lower legs of both experimental group and control group.And the full abbreviation of the above sequence：iterative decomposition of water and fat with echo asymmetry and least-squares estimation (IDEAL) - intelligent quantification (IQ)
Magnetic resonance examination with ultrashort echo time to imaging musculoskeletal ：UTE | 12 months
  All MRI imaging was performed on a clinical 3.0 T General Electric(GE) MR scanner on the lumbar spine and lower legs of both experimental group and control group. And the full abbreviation of the above sequence: ultrashort echo time (UTE)
Magnetic resonance examination for bone morphological observation: ZTE | 12 months
  All MRI imaging was performed on a clinical 3.0 T General Electric(GE) MR scanner on the lower legs of both experimental group and control group.And the full abbreviation of the above sequence: Zero-Echo Time(ZTE)
Magnetic resonance examination to measure changes in the relaxation rate of muscles and blood vessels: SWI | 12 months
  All MRI imaging was performed on a clinical 3.0 T General Electric(GE) MR scanner on the lower legs of both experimental group and control group. And the full abbreviation of the above sequence: Susceptibility-weighted Imaging(SWI)
Bone mineral density（BMD）measured by DXA | 12 months
  The dual energy x-ray absorptiometry (DXA) was performed on the lumbar spine of both experimental group and control group.
Blood biochemistry ：Routine blood was used to detect anemia | 12 months
  Routine blood samples were collected from individuals in the experimental group
Blood biochemistry ：renal function was used for staging CKD | 12 months
  Renal function samples were collected from individuals in the experimental group and control group
Blood biochemistry ：Serum electrolyte was used to detect electrolyte changes | 12 months
  Serum electrolyte samples were collected from individuals in the experimental group
Blood biochemistry ：the ALP、PTH、25-OH VitD、osteocalcin、T-P1NP and β-CTX were used to detect bone metabolism | 12 months
  The above serum samples were collected from individuals in the experimental group
Blood biochemistry ： blood glucose was used to determine the presence or absence of diabetes | 12 months
  Blood glucose samples were collected from individuals in the experimental group
Blood biochemistry ：CK(Creatine kinase) was used to detect muscle lesions | 12 months
  CK samples were collected from individuals in the experimental group
The urine routine was examined to determine whether individuals in the control group and the experimental group had hematuria and proteinuria | 12 months
  The Routine urine samples were collected from individuals in the experimental group and control group

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No